CLINICAL TRIAL: NCT04919200
Title: Measurement of the Total Lung Volume Using Optimized Single-breath Helium Dilution Method in Patients With Obstructive Lung Disease
Brief Title: Optimized Single-breath Helium Lung Volume in Obstructive Lung Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0547
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Obstructive Lung Disease
Keywords: obstructive lung disease; total lung capacity; the single-breath helium dilution; Whole-body plethysmography; correction equation
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Plethysmography, Whole Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- modeling group: Of these 628 individuals, we set 407 patients enrolled from January 2018 to November 2019 as the modeling group
  Interventions: Diagnostic Test: the single-breath helium dilution method and Whole-body plethysmography
- verification cohort: 221 patients enrolled from December 2019-December 2020 served as a prospective verification cohort
  Interventions: Diagnostic Test: the single-breath helium dilution method and Whole-body plethysmography

INTERVENTIONS:
Diagnostic Test: the single-breath helium dilution method and Whole-body plethysmography — The patients with obstructive lung disease simultaneously subjected to the single-breath helium dilution method and Whole-body plethysmography tests.

SUMMARY:
Whole-body plethysmography (WBP) is the gold standard for measuring lung volume, but its clinical application is limited because it requires expensive equipment and is complicated to use. Studies have shown that the single-breath helium dilution (SBHD) method, which is commonly used in clinical practice, significantly underestimates lung volume in patients with obstructive lung disease (OLD). Therefore, by comparing the differences in lung volume measured by the SBHD method and WBP in patients with different severities of obstructive lung disease, we aim to establish a correction equation for the SBHD method to determine the total lung volume in obstructive lung disease patients.

ELIGIBILITY:
Inclusion Criteria:

(1) age 18-80 years and (2) in line with the ATS/ERS definition of obstructive lung disease.

Exclusion Criteria:

(1) contraindications for spirometry, pulmonary diffusion function test, and WBP and (2) history of lung surgery and recent history of chest trauma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 628 patients with obstructive lung disease simultaneously subjected to the single-breath helium dilution method and Whole-body plethysmography tests in Second Affiliated Hospital of Zhejiang University School of Medicine were continuously enrolled from January 2018 to December 2020
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Establishment of the TLC-SBHD correction equation | 2 year
  TLC-adjusted SBHD (L) = -0.669 + 0.756 × TLC-SBHD (L) - 0.047 × FEV1/FVC + 0.039 × height (cm) - 0.009 × weight (kg) (r2 = 0.753 and adjusted r2 = 0.751)

CONTACTS AND LOCATIONS:
Locations (1):
- Key Laboratory of Respiratory Disease of Zhejiang Province, Department of Respiratory and Critical Care Medicine, Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China